CLINICAL TRIAL: NCT01720459
Title: Effects of Micronized Trans-resveratrol Treatment on Clinical, Endocrine, Metabolic and Biochemical Parameters of Women With Polycystic Ovary Syndrome: Placebo-controlled Randomized Single-blind Study
Brief Title: Effects of Micronized Trans-resveratrol Treatment on Polycystic Ovary Syndrome (PCOS) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Beata Banaszewska, MD PhD, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 681/10
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micronized trans-resveratrol (Active Comparator): Micronized trans-resveratrol
  Interventions: Dietary Supplement: Micronized trans-resveratrol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Micronized trans-resveratrol
  Other Names: Micronized trans-resveratrol 500 (Rev Genetics LLC - Miami, FL, USA)
  Arms: Micronized trans-resveratrol
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether micronized trans-resveratrol improves clinical (excessive hair, menstrual cycle), endocrine (androgens)and metabolic (lipids, markers of systemic inflammation) in women with polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

* PCO - Androgen Excess Society criteria: hyperandrogenism (hirsutism) / hyperandrogenemia (testosterone >70ng/dl) and/or oligomenorrhea (<8 spontaneous menses per year) and/or polycystic ovarian morphology on ultrasound
* Normal prolactin, TSH, 17-OH progesterone
* No evidence of androgen producing malignancy, Cushing's syndrome or acromegaly
* Age 18-40

Exclusion Criteria:

* Use of oral contraceptives and/or other steroid hormones 3 months prior to the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
testosterone serum concentration | 3 month therapy

CONTACTS AND LOCATIONS:
Overall Officials: Leszek A Pawelczyk, MD PhD, Study Chair — Poznan University of Medical Sciences; Antoni J Duleba, MD, Study Director — University of California, Davis
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

REFERENCES:
- [Derived] Banaszewska B, Wrotynska-Barczynska J, Spaczynski RZ, Pawelczyk L, Duleba AJ. Effects of Resveratrol on Polycystic Ovary Syndrome: A Double-blind, Randomized, Placebo-controlled Trial. J Clin Endocrinol Metab. 2016 Nov;101(11):4322-4328. doi: 10.1210/jc.2016-1858. Epub 2016 Oct 18. PMID 27754722